CLINICAL TRIAL: NCT03317613
Title: Clinical Trial Assessing the Efficacy of Capsaicin Patch (Qutenza®) in Cancer Patients With Neuropathic Pain
Acronym: CAPSONCO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Institut de Cancérologie de la Loire (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0304; 2017-002476-11 (EudraCT Number)
Record Dates: First submitted 2017-09-21; First posted 2017-10-23 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Neuropathic Pain
Keywords: Neuropathic Pain; Qutenza; Capsaicin; Cancer patient
MeSH Terms: conditions — Neuralgia | interventions — Capsaicin

STUDY DESIGN:
Intervention Model Description: Cancer patients treated with qutenza (capsaicin patch)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Capsaicin (Experimental): Cancer patients presenting neuropathic pain secondary to their anti cancer treatments will receive patch of capsaicin (qutenza) on the painful zones..
  Interventions: Drug: Qutenza

INTERVENTIONS:
Drug: Qutenza — Patients suffering from neuropathic pain will receive patch of capsaicin (qutenza) on the painful zones. Three months after the first application, patients will be allowed to receive another patch if necessary. They will be able to receive one every three months. They will be followed in the study during one year after the first patch application.
  Other Names: 8% capsaicin patch

SUMMARY:
In the oncology area, neuropathic pains are relatively frequent and can be induced by surgery, radiotherapy, or chemotherapy. In usual practice, some units are using qutenza in order to reduce neuropathic pain even though using of this patch for a population of cancer patients has never been demonstrated so far in a prospective study. The present prospective study proposes to evaluate the qutenza efficacy in peripheric neuropathic pain in cancer patients.

DETAILED DESCRIPTION:
Drugs for neuropathic pains are generally represented by antidepressants, anti-epileptics, opioids, lidocaine patch. However, these drugs can frequently be insufficient, and/or can lead to side effects. Qutenza (8% capsaicin patch) presents an interesting alternative.

Qutenza efficacy has been shown in five principal studies conducted on 1988 adults affected by moderate or severe neuropathic pains. All patients presented Postherpetic neuralgia, or HIV associated therapy, or painful diabetic peripheric neuropathies. These studies led to qutenza approbation in Europe and in States in 2009.

In oncology, neuropathic pains are relatively frequent and can be induced by the three big actors of the anti-cancerous therapeutic arsenal (surgery, radiotherapy, chemotherapy). In usual practice, some units are usually using qutenza, but the use of this patch for this kind of patients has not been shown in a prospective study. Advantages of this treatment are numerous, and results presented in other therapeutic area are encouraging its use in oncology.

The present prospective study proposes to evaluate the qutenza efficacy in peripheric neuropathic pain in cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient with at least 18 years old;
* Patient presenting neuropathic pain secondary to an anti-cancerous treatment;
* Patient presenting a DN4 (Neuropathic Pain in Four Questions) score superior or equal to 4 out of 10
* Patient presenting a skin without lesion at the painful area
* Informed consent form signed;
* Patient affiliated to a social security scheme.

Exclusion Criteria:

* Hypersensitivity known to capsaicin;
* Instable or uncontrolled hypertension;
* Painful area localised next to eyes;
* Pregnant or breastfeeding woman;
* Protected people.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Percentage of responders to capsaicin | One month
  Percentage of responders to capsaicin at one month after the first patch application will be calculated with a relief scale completed by patients.

SECONDARY OUTCOMES:
Maximum value of relief | Three months
  Maximum value of relief will be calculated for patients with relief scale completed by patients at three months after the patch application.
Correlation coefficient between the relief score and time before first relief | Three months
  Correlation coefficient between maximal value of relief and time between the beginning of painful signs and first patch application.
Neuropathic pain intensity reported on visual analog scale | One year
  Minimal, average, and maximal values of neuropathic pain reported on visual analog scale will be evaluated.
Number of toxicities reported | One year
  Capsaicin patch induced toxicities will be reported, and quoted according to CTCAE version 4.4.
Number of days of response | One year
  Number of days of response reported by patients where patch are efficient will be reported
Number of days of response to qutenza | One year
  Number of days between the patch set and the apparition of the first effect on patients will be reported.
Size of painful zones | One year
  Size of painful zones will be reported.
Number of prescribed antalgics | One year
  Number of prescribed antalgics will be reported for each patient.
Percentage of patients with a reported chemotherapy | One year
  Percentage of patients with an obligation to report their chemotherapy because of the pain will be calculated.
Percentage of patients who have received at least 75% of the chemotherapy prescribed | One year
  Percentage of patients who have received at least 75% of the chemotherapy prescribed will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie Morisson, MD, Principal Investigator — Institut de Cancérologie Lucien Neuwirth
Locations (3):
- France (3):
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Hospitalier Emile Roux, Le Puy-en-Velay
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez

IPD SHARING:
Plan to Share IPD: No